CLINICAL TRIAL: NCT02183038
Title: Double-blind Study to Compare Efficacy and Safety of Meloxicam 7.5 mg and 15 mg vs. Naproxen Sodium 1100 mg in the Symptomatic Treatment of Acute Non Bacterial Pharyngitis or Pharyngo-tonsillitis Over a Period of 5 Days
Brief Title: Efficacy and Safety of Meloxicam vs. Naproxen Sodium in Patients With Acute Non Bacterial Pharyngitis or Pharyngo-tonsillitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 107.193
Record Dates: First submitted 2014-07-04; First posted 2014-07-08 (Estimated); Last update posted 2014-07-08 (Estimated); Status verified 2014-07

CONDITIONS: Pharyngitis
MeSH Terms: conditions — Pharyngitis | interventions — Naproxen

ARMS (3):
- Meloxicam low & Placebo (Experimental)
  Interventions: Drug: Meloxicam low; Drug: Meloxicam placebo high; Drug: Naproxen sodium placebo
- Meloxicam high & Placebo (Experimental)
  Interventions: Drug: Meloxicam high; Drug: Meloxicam placebo low; Drug: Naproxen sodium placebo
- Naproxen sodium & Placebo (Active Comparator)
  Interventions: Drug: Naproxen sodium; Drug: Meloxicam placebo low; Drug: Meloxicam placebo high

INTERVENTIONS:
Drug: Meloxicam low
  Arms: Meloxicam low & Placebo
Drug: Meloxicam high
  Arms: Meloxicam high & Placebo
Drug: Naproxen sodium
  Arms: Naproxen sodium & Placebo
Drug: Meloxicam placebo low
  Arms: Meloxicam high & Placebo; Naproxen sodium & Placebo
Drug: Meloxicam placebo high
  Arms: Meloxicam low & Placebo; Naproxen sodium & Placebo
Drug: Naproxen sodium placebo
  Arms: Meloxicam high & Placebo; Meloxicam low & Placebo

SUMMARY:
Study to assess the efficacy and tolerability of Meloxicam once daily dose of 7.5 mg and 15 mg compared with 1100 mg of naproxen sodium in the symptomatic treatment of acute non bacterial pharyngitis or pharyngo-tonsillitis, over a period of 5 days.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 18 years or above
* Ambulatory patients
* Start of symptoms within the previous 24 hours
* Patients suffering from acute non bacterial pharyngitis or pharyngo-tonsillitis diagnostic, under the following criteria:

  * spontaneous pharyngeal pain presence greater than 35 mm on a 100 mm visual analog scale (VAS)
  * Pharyngeal pain presence on swallowing greater than 35 mm on a 100 mm VAS
  * Pharyngeal and/or amygdaline hyperemia
  * Absence of purulent plaques
  * Negative test for β-haemolytic Streptococcus on pharyngeal exudate
* Therapy with NSAID (Non-Steroid Anti-Inflammatory Drug) is required or recommended
* Patient's informed consent in accordance with local law and ICH GCP (International Conference of Harmonization Good Clinical Practice) , before inclusion into the the trial

Exclusion Criteria:

* Suspicion of acute pharyngitis or pharyngo-tonsillitis from bacterial origin by clinical criteria; Several impairment of patients condition, indicated by one or more or the following symptoms:

  * Extremely rapid onset of clinical picture
  * Very high fever (>38.5°C)
  * Severe pharyngeal pain
  * Cervical adenopathy
  * Intense headache
  * Purulent pharyngeal plaques, evidence of peritonsillar abscess or phlegmon
* Known or suspected hypersensitivity to the trial drug or NSAIDs
* Positive test for β-haemolytic Streptococcus on pharyngeal exudate
* Therapy with antimicrobial agents prior to start of the trial
* Chronic infections
* Infectious mononucleosis
* Active peptic ulcer within the past 6 months
* Pregnancy or breast feeding precaution: attention should be drawn to reports that NSAIDs were reported to decrease the efficacy of intrauterine devices
* Asthma, nasal polyps, angioneurotic edema or urticaria following the administration of aspirin or NSAIDs
* Concomitant treatment with anti-coagulants (including heparin), lithium or methotrexate
* Concomitant administration of other NSAIDs (including high-dose > 1500 mg at day aspirin) or analgesic agents
* Administration of any NSAID during the last three days or analgesics 6 hours prior to the first administration of the trial drug
* Present treatment or treatment within the last two months with corticosteroids
* Historically know of impaired renal function (serum urea > 125 % of the upper limit of normal range; serum creatinine > 150 % of the upper limit of normal range)
* Historically know of severe liver injury (alanine amino transferase ALAT > 2 x the upper normal range limit or aspartate amino transferase ASAT > 2 x the upper normal range limit)
* Historically know of hematological disorder (platelet count < 100,000/mm3, leucocyte count < 3,000/mm3)
* Participation in another clinical trial during this study or during the previous month
* Previous participation in this trial
* Patient unable to comply with the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 390 (Actual)
Dates: Start 1998-07; Primary Completion 1999-02 (Actual)

PRIMARY OUTCOMES:
Change in intensity of spontaneous pharyngeal pain | Baseline, day 3 and 5
Change in intensity of pharyngeal pain on swallowing | Baseline, day 3 and 5

SECONDARY OUTCOMES:
Final global assessment of efficacy by patient | Day 5
Final global assessment of efficacy by investigator | Day 5
Final global assessment of tolerability by patient | Day 5
Final global assessment of tolerability by investigator | Day 5
Occurrence of disease systemic manifestations (fever, and general malaise) | up to 5 days
Occurrence of pharyngeal hyperemia | up to 5 days
Assessment of patient status | Day 5
Occurrence of treatment withdrawal due to lack of efficacy | up to 5 days
Occurrence of perforation, ulceration, bleeding (PUB) of the upper gastro-intestinal tract (stomach or duodenum) | up to day 5
Intensity of adverse events | up to 19 days
Number of patients who withdraw due to adverse event | up to 19 days
Incidence of significant laboratory adverse events | up to 19 days
Occurrence and duration of hospital stay due to Gastro-Intestinal Serious Adverse Events (GI-SAE) | up to 19 days
Occurrence and duration of hospital stay due to adverse events related to trial drug administration | up to 19 days
Occurrence of an additional visit at physician due to gastro-intestinal adverse event (GI-AE) | up to 19 days
Number of patients with adverse events | up to 19 days
Number of patients with adverse events related to trial drug | up to 19 days